CLINICAL TRIAL: NCT02416453
Title: A Randomized, Observer-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability and Immunogenicity of Three Prime-Boost Regimens of the Candidate Prophylactic Vaccines for Ebola Ad26.ZEBOV and MVA-BN-Filo in Healthy Adults in Europe
Brief Title: A Study to Assess Safety, Tolerability, and Immunogenicity of Three Heterologus 2-dose Regimens of the Candidate Prophylactic Vaccines for Ebola in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR107227; VAC52150EBL2001 (Other: Janssen Vaccines & Prevention B.V.); 2015-000596-27 (EudraCT Number)
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Ebola Viral Disease
Keywords: Healthy; Ebola viruses; Ebola Viral Disease (EVD); Filoviruses; Monovalent vaccine; Human adenovirus serotype 26 (Ad26) encoding the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN Filo); Safety; Immunogenicity; Inserm and University of Oxford

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive intramuscular (IM) injection of Ad26.ZEBOV/Placebo on Day 1 followed by IM injection of MVA-BN-Filo/Placebo on Day 29.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo
- Group 2 (Experimental): Participants will receive IM injection of Ad26.ZEBOV/Placebo on Day 1 followed by IM injection of MVA-BN-Filo/Placebo on Day 57.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo
- Group 3 (Experimental): Participants will receive IM injection of Ad26.ZEBOV/Placebo on Day 1 followed by IM injection of MVA-BN-Filo/Placebo on Day 85.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo

INTERVENTIONS:
Biological: MVA-BN-Filo — One 0.5 mL intramuscular (IM) injection of 1E8 Infectious Unit [Inf. U.] on Day 29, 57, or 85.
Biological: Ad26.ZEBOV — One 0.5 mL IM injection of 5E10 viral particles (vp) on Day 1.
Biological: Placebo — One 0.5 mL IM injection of 0.9% saline on Day 1 and Day 29, 57, or 85.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of 3 vaccination schedules of Ad26.ZEBOV and MVA-BN-Filo administered intramuscularly (IM) as 2-dose heterologous regimens.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, placebo-controlled, parallel-group, multicenter, Phase 2 study evaluating the safety, tolerability and immunogenicity of 2-dose heterologous regimens using Ad26.ZEBOV and MVA-BN-Filo administered to healthy adults participants in Europe. The study involves a screening period of up to 12 weeks, a vaccination period in which participants will be vaccinated with Ad26.ZEBOV (dose 1) followed by vaccination with MVA-BN-Filo (dose 2) 28, 56 or 84 days later, and a post-vaccination phase until 6 months post dose 2 visit (Days 209, 237 or 265). After unblinding, only participants who received Ad26.ZEBOV and/or MVA-BN-Filo will continue the study until the Day 365 visit (or until the start of the roll-over study or for an additional 12 months [whichever comes first] for participants in France who agree to continue the long-term follow-up after Day 365) to assess long-term safety and immunogenicity. Participants will enroll into 3 cohorts: that is, Cohort 1 (Participants will receive Ad26.ZEBOV and MVA-BN-Filo in an open-label fashion), Cohort 2 (Participants will be randomized to receive the 2-dose heterologous vaccine regimen with either Ad26.ZEBOV followed by MVA-BN-Filo, or placebo in a 14:1 ratio) and Cohort 3 (Participants will be randomized to receive the 2-dose heterologous vaccine regimen with either Ad26.ZEBOV followed by MVA-BN-Filo, or placebo in a 10:3 ratio). In Cohorts 2 and 3, core immunogenicity assessments (humoral and cellular assays) will be performed. In Cohort 2, additional immunogenicity assessments will be done. In Cohort 1, plasma blast response kinetics will be evaluated. Safety will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy in the Investigator's clinical judgment on the basis of medical history, physical examination, electrocardiogram (ECG) and vital signs performed at Screening
* Must be healthy on the basis of clinical laboratory tests performed at Screening. If the results of the laboratory screening tests are outside the normal reference ranges, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study
* Before randomization, a woman must be either of childbearing potential and practicing (or intending to practice) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies, beginning at least 28 days prior to vaccination OR not of childbearing potential: postmenopausal (greater than [>] 45 years of age with amenorrhea for at least 2 years or lesser than or equal to [<=] 45 years of age with amenorrhea for at least 6 months, and a serum follicle stimulating hormone (FSH) level >40 international unit per milliliter [IU/L]); permanently sterilized (for example, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* Woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at Screening and a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* Man who is sexually active with a woman of childbearing potential and has not had a vasectomy performed more than 1 year prior to screening must be willing to use condoms for sexual intercourse beginning prior to enrollment

Exclusion Criteria:

* Having received any candidate Ebola vaccine
* Diagnosed with Ebola virus disease, or prior exposure to Ebola virus, including travel to West Africa less than 1 month prior to screening. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone
* Having received any experimental candidate adenovirus serotype 26 (vector: Ad26) or Modified Vaccinia Ankara (MVA-) based vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines including known allergy to egg, egg products and aminoglycosides
* Presence of acute illness or temperature greater than or equal to 38.0 C on Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.; Inserm Clinical Trials, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (11):
- France (8):
  - Créteil
  - Marseille
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Etienne
  - Strasbourg
  - Tours
- United Kingdom (3):
  - London
  - Oxford
  - Southampton

REFERENCES:
- [Derived] Lacabaratz C, Durand M, Wiedemann A, Foucat E, Surenaud M, Krief C, Guillaumat L, Robinson C, Luhn K, Bockstal V, Thiebaut R, Richert L, Levy Y. Innate and Cellular Immune Response to the Ebola Vaccine Ad26.ZEBOV, MVA-BN-Filo: An Ancillary Study of the EBL2001 Phase 2 Trial. J Infect Dis. 2025 Feb 4;231(1):230-240. doi: 10.1093/infdis/jiae360. PMID 39012798
- [Derived] Barry H, Lhomme E, Surenaud M, Nouctara M, Robinson C, Bockstal V, Valea I, Somda S, Tinto H, Meda N, Greenwood B, Thiebaut R, Lacabaratz C. Helminth exposure and immune response to the two-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen. PLoS Negl Trop Dis. 2024 Apr 11;18(4):e0011500. doi: 10.1371/journal.pntd.0011500. eCollection 2024 Apr. PMID 38603720
- [Derived] Pollard AJ, Launay O, Lelievre JD, Lacabaratz C, Grande S, Goldstein N, Robinson C, Gaddah A, Bockstal V, Wiedemann A, Leyssen M, Luhn K, Richert L, Betard C, Gibani MM, Clutterbuck EA, Snape MD, Levy Y, Douoguih M, Thiebaut R; EBOVAC2 EBL2001 study group. Safety and immunogenicity of a two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in adults in Europe (EBOVAC2): a randomised, observer-blind, participant-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2021 Apr;21(4):493-506. doi: 10.1016/S1473-3099(20)30476-X. Epub 2020 Nov 17. PMID 33217361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 423 participants were randomized (408 participants in Groups 1 to 3 and 15 participants in Group 4). Among them, 421 participants received at least one dose of study vaccines. Two participants were randomized but not vaccinated.
Groups:
- Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval): Participants received intramuscular (IM) injection of Ad26.ZEBOV at 5*10^10 viral particles (vp) as dose 1 on Day 1 followed by IM injection of MVA-BN-filo at 1*10^8 infectious units (Inf.U) (nominal titer) as dose 2 on Day 29.
- Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval); Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval): Participants received IM injection of Ad26.ZEBOV at 5*10^10 vp as dose 1 on Day 1 followed by IM injection of MVA-BN-filo at 1*10^8 Inf.U (nominal titer) as dose 2 on Day 57.
- Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval); Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval): Participants received IM injection of Ad26.ZEBOV at 5*10^10 vp as dose 1 on Day 1 followed by IM injection of MVA-BN-filo at 1*10^8 Inf.U (nominal titer) as dose 2 on Day 85.
- Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval): Participants received IM injection of Ad26.ZEBOV at 5*10^10 vp as dose 1 on Day 1 followed by IM injection of MVA-BN-filo at 1*10^8 Inf.U (nominal titer) as dose 2 on Day 29.
- Group 1: Pooled Cohorts II and III: Placebo: Participants received IM injection of placebo on Day 1 and Day 29.
- Group 2: Pooled Cohorts II and III: Placebo: Participants received IM injection of placebo on Day 1 and Day 57.
- Group 3: Pooled Cohorts II and III: Placebo: Participants received IM injection of placebo on Day 1 and Day 85.
- Group 4: Ad26.ZEBOV: Participants received IM injection of Ad26.ZEBOV at 5*10^10 vp on Day 1.
- Group 4: Placebo: Participants received IM injection of placebo Day 1.
Period: Overall Study
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo | Group 4: Ad26.ZEBOV | Group 4: Placebo
Started | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18 | 13 | 2
Completed | 7 | 7 | 9 | 97 | 12 | 98 | 11 | 94 | 13 | 13 | 2
Not Completed | 3 | 3 | 1 | 15 | 1 | 16 | 2 | 12 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 8 | 0 | 5 | 1 | 3 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 5 | 1 | 8 | 0 | 8 | 4 | 0 | 0
Not completed — PARTICIPANT UNABLE TO ATTEND ANY FURTHER | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PARTICIPANT HAS MOVED TO SINGAPORE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo | Group 4: Ad26.ZEBOV | Group 4: Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18 | 13 | 2 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (12.95) | 47.4 (16.53) | 38.7 (13.99) | 41 (15) | 39.1 (13.9) | 41 (14.02) | 38.2 (13.66) | 38.3 (14.34) | 41.1 (15.11) | 37.9 (11.37) | 47 (4.24) | 40 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 57 | 6 | 62 | 8 | 53 | 10 | 3 | 1 | 217
  Male | 6 | 4 | 3 | 55 | 7 | 52 | 5 | 53 | 8 | 10 | 1 | 204
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 0 | 3 | 1 | 5 | 1 | 0 | 0 | 13
  Black or African American | 0 | 0 | 2 | 10 | 1 | 8 | 2 | 9 | 1 | 3 | 0 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 8 | 97 | 12 | 102 | 10 | 89 | 16 | 10 | 2 | 365
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 0 | 0 | 54 | 7 | 55 | 7 | 50 | 9 | 13 | 2 | 197
  United Kingdom | 10 | 10 | 10 | 58 | 6 | 59 | 6 | 56 | 9 | 0 | 0 | 224

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unsolicited Adverse Events (Groups 1, 2 and 3)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, it does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal product. Unsolicited adverse events were events which were reported by the participant voluntarily or obtained by means of interviewing the participant in a nondirected manner at study visits.
Time Frame: Up to 42-day post dose 2 visit (Day 1 to Day 127)
Population: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo), regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18
Participants | 4 | 6 | 6 | 62 | 6 | 52 | 7 | 46 | 8

2. Primary Outcome: Number of Participants With Serious Adverse Events (Groups 1, 2 and 3)
Description: A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18
Participants | 0 | 1 | 0 | 2 | 0 | 4 | 1 | 5 | 1

3. Primary Outcome: Number of Participants With Immediate Reportable Events (Groups 1, 2 and 3)
Description: The following neuroinflammatory disorders were considered immediate reportable events and which had to be reported to the sponsor within 24 hours of becoming aware of the event. Neuroinflammatory disorders included: cranial nerve disorders including paralyses/paresis (example: bell's palsy), optic neuritis, multiple sclerosis, transverse myelitis, guillain-barre syndrome including miller fisher syndrome, bickerstaff's encephalitis and other variants, acute disseminated encephalomyelitis, including site-specific variants (example: non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis), myasthenia gravis and lambert-eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, including chronic inflammatory, demyelinating polyneuropathy, multifocal motor neuropathy, and polyneuropathies associated with monoclonal gammopathy, narcolepsy, isolated paresthesia of more than 7 days duration.
Time Frame: Up to Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0

4. Primary Outcome: Number of Participants With Solicited Local Adverse Events (Groups 1, 2 and 3)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post first vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site.
Time Frame: 7 days post-dose 1 (Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18
Participants | 8 | 6 | 8 | 63 | 3 | 65 | 2 | 78 | 4

5. Primary Outcome: Number of Participants With Solicited Local Adverse Events (Groups 1, 2 and 3)
Description: as for outcome 4
Time Frame: 7 days post-dose 2 (Up to Day 92)
Population: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo), regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 8 | 9 | 9 | 91 | 10 | 83 | 7 | 62 | 11
Participants | 4 | 5 | 8 | 46 | 2 | 49 | 0 | 41 | 0

6. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (Groups 1, 2 and 3)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Time Frame: 7 days post-dose 1 (Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 112 | 13 | 114 | 13 | 106 | 18
Participants | 8 | 10 | 10 | 89 | 7 | 84 | 8 | 82 | 7

7. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (Groups 1, 2 and 3)
Description: as for outcome 6
Time Frame: 7 days post-dose 2 (Up to Day 92)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 8 | 9 | 9 | 91 | 10 | 83 | 7 | 62 | 11
Participants | 6 | 5 | 5 | 42 | 5 | 36 | 2 | 38 | 4

8. Secondary Outcome: Number of Participants With Unsolicited Adverse Events (Group 4)
Description: An AE is any untoward medical occurrence in a clinical study subject administered a medicinal product, it does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal product. Unsolicited adverse events were events which were reported by the participant voluntarily or obtained by means of interviewing the participant in a nondirected manner at study visits.
Time Frame: Up to 28-day post dose 1 (Day 29)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.ZEBOV | Group 4: Placebo
Number analyzed (Participants) | 13 | 2
Participants | 6 | 1

9. Secondary Outcome: Number of Participants With Serious Adverse Events (Group 4)
Description: A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.ZEBOV | Group 4: Placebo
Number analyzed (Participants) | 13 | 2
Participants | 2 | 0

10. Secondary Outcome: Number of Participants With Immediate Reportable Events (Group 4)
Description: The following neuroinflammatory disorders were considered immediate reportable events which had to be reported to the sponsor within 24 hours of becoming aware of the event. Neuroinflammatory disorders included: cranial nerve disorders including paralyses/paresis (example: bell's palsy), optic neuritis, multiple sclerosis, transverse myelitis, guillain-barre syndrome including miller fisher syndrome, bickerstaff's encephalitis and other variants, acute disseminated encephalomyelitis, including site-specific variants (example: non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis), myasthenia gravis and lambert-eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, including chronic inflammatory, demyelinating polyneuropathy, multifocal motor neuropathy, and polyneuropathies associated with monoclonal gammopathy, narcolepsy, isolated paresthesia of more than 7 days duration.
Time Frame: Up to Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.ZEBOV | Group 4: Placebo
Number analyzed (Participants) | 13 | 2
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (Group 4)
Description: as for outcome 4
Time Frame: 7 days after each vaccination (Up to Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.ZEBOV | Group 4: Placebo
Number analyzed (Participants) | 13 | 2
Participants | 8 | 0

12. Secondary Outcome: Number of Participants With Solicited Systemic Adverse Events (Group 4)
Description: as for outcome 6
Time Frame: 7 days after each vaccination (Up to Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.ZEBOV | Group 4: Placebo
Number analyzed (Participants) | 13 | 2
Participants | 11 | 1

13. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against Ebola Virus Glycoprotein (EBOV GP) Measured Using Filovirus Animal Non-Clinical Group (FANG) Enzyme-linked Immunosorbent Assay (ELISA) (Groups 1, 2 and 3)
Description: GMCs of antibodies binding to EBOV GP using FANG ELISA were reported and were measured in ELISA unit per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using FANG ELISA to determine humoral responses following vaccination. For ELISA binding antibody responses, values below the lower limit of quantification (LLOQ) (36.11 ELISA units/mL). The outcome measure was planned to be reported at 21-day post dose 2. Therefore, the results are reported for Group 1, 2 and 3 only.
Time Frame: At 21-days post dose 2 (Day 50 for Group 1; Day 78 for Group 2; and Day 106 for Group 3)
Population: The per protocol analysis set included all randomized and vaccinated participants, who received both the prime and boost vaccinations (administered within the protocol-defined window), have at least 1 post-vaccination (that is, after the date of vaccination) evaluable immunogenicity sample, and have no major protocol violations influencing the immune response. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo
Number analyzed (Participants) | 77 | 7 | 69 | 7 | 48 | 6
EU/mL | 4627 [3649 to 5867] | NA [NA to 55] — Here, 'NA' signifies that Geometric mean and lower limit of 95% CI were not calculated because post dose values were less than LLOQ (36.11 ELISA units/mL). | 10131 [8554 to 11999] | NA [NA to NA] — Here, 'NA' signifies that Geometric mean and CI were not calculated because post dose values were less than LLOQ (36.11 ELISA units/mL). | 11312 [9072 to 14106] | NA [NA to NA] — Here, 'NA' signifies that Geometric mean and CI were not calculated because post dose values were less than LLOQ (36.11 ELISA units/mL).

ADVERSE EVENTS:
Time Frame: Up to Day 365
Description: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo), regardless of the occurrence of protocol deviations.
Arm/Group | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) | Group 1: Pooled Cohorts II and III: Placebo | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) | Group 2: Pooled Cohorts II and III: Placebo | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) | Group 3: Pooled Cohorts II and III: Placebo | Group 4: Ad26.ZEBOV | Group 4: Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/112 | 0/13 | 0/114 | 0/13 | 0/106 | 0/18 | 0/13 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 2/112 | 0/13 | 4/114 | 1/13 | 5/106 | 1/18 | 2/13 | 0/2
Other Adverse Events (participants affected / at risk) | 4/10 | 5/10 | 6/10 | 41/112 | 6/13 | 30/114 | 7/13 | 26/106 | 8/18 | 6/13 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) (N=10) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) (N=10) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) (N=10) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) (N=112) | Group 1: Pooled Cohorts II and III: Placebo (N=13) | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) (N=114) | Group 2: Pooled Cohorts II and III: Placebo (N=13) | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) (N=106) | Group 3: Pooled Cohorts II and III: Placebo (N=18) | Group 4: Ad26.ZEBOV (N=13) | Group 4: Placebo (N=2)
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Human papilloma virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Miller Fisher syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small fibre neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) (N=10) | Group 2: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) (N=10) | Group 3: Cohort I: Ad26.ZEBOV, MVA-BN-Filo (84-Day Interval) (N=10) | Group 1: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (28-Day Interval) (N=112) | Group 1: Pooled Cohorts II and III: Placebo (N=13) | Group 2: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo (56-Day Interval) (N=114) | Group 2: Pooled Cohorts II and III: Placebo (N=13) | Group 3: Pooled Cohorts II and III: Ad26.ZEBOV, MVA-BN-Filo, (84-Day Interval) (N=106) | Group 3: Pooled Cohorts II and III: Placebo (N=18) | Group 4: Ad26.ZEBOV (N=13) | Group 4: Placebo (N=2)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 7 | 0 | 6 | 0 | 3 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 6 | 1 | 6 | 1 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 3 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 3 | 0 | 2 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 5 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 3 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02416453/SAP_000.pdf
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT02416453/Prot_001.pdf